CLINICAL TRIAL: NCT04215055
Title: Comparative Evaluation Between the Effectiveness of Vibration Assisted Syringe and Conventional Syringe in Decreasing Children Pain and Anxiety Perception During Local Anesthetic Injection ) Randomized Controlled Clinical Trial (
Brief Title: Comparative Evaluation Between the Effectiveness of Vibration Assisted Syringe and Conventional Syringe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdallah Mohamed Abdallah, dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vibraject in Dentistry
Record Dates: First submitted 2019-12-26; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Anxiety, Dental
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): Group I (study group); children receiving intraoral injection of local anasethia using the vibration assisted syringe.
  Interventions: Device: vibraject
- control group (Active Comparator): Group II (control group): children receiving intraoral injection of local anasethia using the standard syringe.
  Interventions: Device: vibraject

INTERVENTIONS:
Device: vibraject — VibraJect; is a small battery-operated attachment that snaps on to the standard dental syringe. It delivers a high-frequency vibration to the needle which is strong enough for the patient to feel.

SUMMARY:
The study will be conducted to evaluate the effect of the vibration assisted syringe on pain perception and anxiety in children during intra oral injection of local anesthesia in comparison with conventional syringe.

DETAILED DESCRIPTION:
As for granted the main concern in pediatric dentistry is to guarantee a positive response from child for any further appointments, that's why we aim to manage a successful dental procedure keeping a stress free situation. Conventional local anesthetic technique is the most commonly used technique for anesthetizing teeth but in turn it has shown the highest levels of discomfort in comparison with other techniques. VibraJect is vibration associated syringe device, it is simple and cost effective solution to alleviate injection discomfort. It works because the light pressure of a Vibraject injection is carried rapidly to the brain by thicker insulated nerve tissues. In contrast, the needle prick travels on thinner nerve tissues, arriving too late for the brain to register the sensation. Vibraject is good news for the patient, because the anesthetic itself causes virtually no discomfort and good news for the dentist, who can work easily knowing that patient, is comfortable.

ELIGIBILITY:
inclusion criteria

1. Cooperative patient. (rating 4 or 3 based on Frankl behavior scale).
2. Children aging from 4 to 6 years
3. Suffering from one or more deep carious lesions in their primary molars.
4. Restorable primary molars

Exclusion Criteria:

1. Medically compromised patients.
2. Uncooperative children (rating 1 or 2 on the Frankl behavior scale) needing special line of treatment through general anesthesia.
3. Signs and symptoms of irreversible pulpitis, spontaneous pain, necrosis or any signs and symptoms of abscess.
4. Presence of any radiographic signs of abscess, bone loss, internal or external root resorption.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 46 (Estimated)
Dates: Start 2020-02-08 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Pain rating scale | baseline
  Visual linear analogue scale

SECONDARY OUTCOMES:
anxiety | baseline
  Visual facial anxiety scale

CONTACTS AND LOCATIONS:
Overall Officials: mohamed abdallah, Principal Investigator — Cairo University

REFERENCES:
- [Background] Roeber B, Wallace DP, Rothe V, Salama F, Allen KD. Evaluation of the effects of the VibraJect attachment on pain in children receiving local anesthesia. Pediatr Dent. 2011 Jan-Feb;33(1):46-50. PMID 21406147
- [Background] Wilson S. Management of child patient behavior: quality of care, fear and anxiety, and the child patient. J Endod. 2013 Mar;39(3 Suppl):S73-7. doi: 10.1016/j.joen.2012.11.040. PMID 23439049